CLINICAL TRIAL: NCT05214495
Title: Efficacy of Topical Oral Omega-3 Hydrogel in Prevention of Radiation-induced Oral Mucositis in Head and Neck Cancer Patients: A Randomized Controlled Clinical Trial
Brief Title: Omega-3 Hydrogel and Prevention of Oral Mucositis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Basma Morsy (Other)
Responsible Party: Sponsor-Investigator, Basma Morsy, Principal Investigator, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0290-09/2021
Record Dates: First submitted 2022-01-02; First posted 2022-01-28 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Mucositis Oral
MeSH Terms: conditions — Stomatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Topical oral Omega-3 hydrogel group (Experimental): Patients will be given topical oral Omega-3 hydrogel
  Interventions: Drug: topical oral Omega-3 hydrogel
- Conventional preventive treatment group (Active Comparator): Patients will be given conventional preventive treatment
  Interventions: Drug: conventional preventive treatment

INTERVENTIONS:
Drug: topical oral Omega-3 hydrogel — Topical oral Omega-3 hydrogel prepared from fish oil
  Arms: Topical oral Omega-3 hydrogel group
Drug: conventional preventive treatment — topical treatment including antifungal agents, anti-inflammatory mouthwash, sodium bicarbonate mouthwash.
  Topical anesthetics agent, topical analgesic gel as well as systemic analgesics (if needed)
  Arms: Conventional preventive treatment group

SUMMARY:
Oral mucositis (OM) is recognized as one of the most frequent debilitating sequela encountered by head and neck cancer (HNC) patients treated by radiotherapy. The objective of the study is to assess primarily the effect of topical oral Omega-3 hydrogel in prevention of radiation-induced oral mucositis and secondarily, to test the effect of topical oral Omega-3 hydrogel on oral microbiome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are going to receive radiotherapy as a treatment of head and neck cancer either as postoperative (adjuvant) therapy or definitive therapy.
2. Patients whose radiotherapy treatment planned dose is 50 Gy or above
3. Males and females with an age not less than 18 years
4. Patients receiving radiotherapy alone or receiving concomitant cisplatin (or carboplatin) with radiotherapy.

Exclusion Criteria:

1. Patients under Anticoagulants such as warfarin, heparin, or aspirin.
2. Patients suffering from any uncontrolled systemic diseases (such as diabetes, cardiovascular, liver disorder, renal dysfunction)
3. Patients with findings of any physical or mental abnormality which would interfere with or be affected by the study procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-02-09 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Oral Mucositis Severity | up to 6 weeks
  Radiation induced head and neck toxicity will be scored by a scale based on clinical features from Common Terminology Criteria for Adverse Events (CTCAE) v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Alexandria University, Alexandria, Egypt